CLINICAL TRIAL: NCT03453723
Title: Pain Prevention During Propofol Infusion in Pediatric: Hypnoanalgesia of the Hand Versus Lidocaine.
Acronym: PROPLIDHYPNO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/17/0041; 2017-002630-22 (EudraCT Number)
Record Dates: First submitted 2018-02-08; First posted 2018-03-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2020-11

CONDITIONS: Pain
Keywords: hypnoanalgesia; lidocaine; propofol; children
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magic glove hypnosis (Experimental): Magic glove hypnosis technique use before propofol infusion
  Interventions: Procedure: Magic glove hypnosis technique
- lidocaine (Active Comparator): extemporaneous mixture with lidocaine for propofol infusion
  Interventions: Drug: lidocaine

INTERVENTIONS:
Procedure: Magic glove hypnosis technique — Realization of the magic glove hypnosis technique by an expert physician trained in hypnosis, according to a classic discourse before : intravenous infusion with 1% propofol (3 mg/kg with 600 ml / h electric syringe pump). Use and dose in accordance with the SPC.
  Arms: magic glove hypnosis
Drug: lidocaine — intravenous infusion with an extemporaneous mixture of 18 volumes 1% propofol (180mg) for 2 volumes of 1% lidocaine (2ml) with 600 ml / h electric syringe pump. Use and dose in accordance with the SPC.
  Arms: lidocaine

SUMMARY:
The simplicity of the implementation and the effectiveness of hypno-analgesia (via the magic glove technique) has already been proven in some research work, during the installation of peripheral venous route. An unpublished preliminary study has shown that this method appears to be the most effective in preventing pain during pediatric propofol injection.

The purpose is to compare the effectiveness of hypno-analgesia of the hand by the "magic glove technique" to lidocaine used in an extemporaneous mixture in the prevention of pain with injection of propofol during intravenous induction in children aged 7 to 14 years

DETAILED DESCRIPTION:
Propofol is a hypnotic of choice, because of its speed of action, its dose-effect relationship (allowing titrated inductions), its anti-emetic effect, as well as its delay and its short duration of action. Among its side effects, the pain during its injection occupies a significant part in pediatrics (60% in adults, up to 85% in children).

It is most often described as an unpleasant sensation, discomfort or even a burn at the point of puncture, going up along the path of the vein and can extend to the whole arm. The mechanism of this pain is still poorly understood at this time. Several mechanisms have been mentioned such as activation of the bradykinin cascade, a direct stimulation of the free nociceptive venous nerve endings.A meta-analysis concludes in adults that the two most effective techniques are a puncture site on the ulnar vein and a pretreatment of the vein by Lidocaine. In children, the anatomical differences, the notion of protection of the venous capital from the first vascular approach, whatever the prognosis of the patient and the competence of the operator will influence the choice of the material, the choice of the site and the puncture technique. Several pediatric studies have attempted to reduce this injection pain by other techniques. A panel of products has been tested with different drug orientations or not. The suggestion centered on analgesia of the hand is a powerful technique, adapted to acute pain. The pain sensation will thus be partially or completely replaced by a sensation of a different nature, thus attenuating the nociceptive process. This technique has not been studied during injection with propofol.

ELIGIBILITY:
Inclusion Criteria:

* Children from 7 to 14 years old.
* Admitted for programmed or ambulatory surgery under general anesthesia.
* ASA I to II. (ASA1: Normal patient or ASA 2: Patient with moderate systemic abnormality).
* Parents or legal guardians who have signed informed consent to the inclusion visit.

Exclusion Criteria:

* Children under 7, over 14
* In regulated girls, presence of a pregnancy
* ASA III, IV
* Contraindication to propofol (known hypersensitivity to propofol or to one of its constituents)
* Contraindications to lidocaine (known hypersensitivity to lidocaine hydrochloride, amide bonded local anesthetics or to any of the excipients, patients with recurrent porphyria)
* Contraindications to nitrous oxide
* Patient whose clinical condition requires titration of propofol during induction, for good hemodynamic tolerance.
* Refusal by the child or the parents of intravenous induction.
* Psychological distress (agitation, mental deficiencies, communication disorders, deafness problems).
* Analgesic or sedative treatment within 24 hours before induction.
* Locoregional or perimedullary anesthesia before anesthetic induction.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Score: Cameron Type Scale | Day 1
  The reactions of the child from the beginning of the injection are filmed by an outside observer.
  At the end of the 3 mg / kg, the observation is stopped. From a distance, a member of the Children's Hospital Pain Unit will blindly display, by viewing child-centered videos, a pain score, according to Cameron's score [0 = No pain ( no reaction); 1 = slight pain (grimace); 2 = Moderate pain (grimaces + cries / moans); 3 = severe pain (crying / crying + hand removal).].
  A score greater than or equal to two represents a significant pain at induction.

SECONDARY OUTCOMES:
Satisfaction assessment | Day 1
  Evaluation of the satisfaction as soon as the child is able to leave the post interventional surveillance room (sspi) by an analog evaluation scale of the degree of satisfaction. A score ≤ 7 expressing dissatisfaction on his part, the reasons for this possible discontent will then be requested. Then, we will ask him, in case he should be asleep, if he wants us to proceed in the same way.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Madeleine Polomeni, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital des enfants - Pôle Anesthésie-Réanimation., Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cameron E, Johnston G, Crofts S, Morton NS. The minimum effective dose of lignocaine to prevent injection pain due to propofol in children. Anaesthesia. 1992 Jul;47(7):604-6. doi: 10.1111/j.1365-2044.1992.tb02335.x. PMID 1626674
- [Background] Jalota L, Kalira V, George E, Shi YY, Hornuss C, Radke O, Pace NL, Apfel CC; Perioperative Clinical Research Core. Prevention of pain on injection of propofol: systematic review and meta-analysis. BMJ. 2011 Mar 15;342:d1110. doi: 10.1136/bmj.d1110. PMID 21406529
- [Background] Nishimoto R, Kashio M, Tominaga M. Propofol-induced pain sensation involves multiple mechanisms in sensory neurons. Pflugers Arch. 2015 Sep;467(9):2011-20. doi: 10.1007/s00424-014-1620-1. Epub 2014 Oct 10. PMID 25301522
- [Background] Depue K, Christopher NC, Raed M, Forbes ML, Besunder J, Reed MD. Efficacy of intravenous lidocaine to reduce pain and distress associated with propofol infusion in pediatric patients during procedural sedation. Pediatr Emerg Care. 2013 Jan;29(1):13-6. doi: 10.1097/PEC.0b013e31827b227e. PMID 23283255
- [Background] Kuttner L. Pediatric hypnosis: pre-, peri-, and post-anesthesia. Paediatr Anaesth. 2012 Jun;22(6):573-7. doi: 10.1111/j.1460-9592.2012.03860.x. PMID 22594409
- [Result] Polomeni MM, Huguet T, Mariotti M, Larcher C, Delort F, Minville V, Kern D. Avoiding pain during propofol injection in pediatric anesthesia: Hypnoanalgesia of the hand versus intravenous lidocaine. Paediatr Anaesth. 2024 Aug;34(8):742-749. doi: 10.1111/pan.14909. Epub 2024 May 2. PMID 38693886